CLINICAL TRIAL: NCT04653233
Title: University of Health Sciences, Hamidiye Nursing Faculty, Istanbul, Turkey
Brief Title: Effectiveness of Haptic Technology in Teaching Urinary Catheterization Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Assistant Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1898
Record Dates: First submitted 2020-11-20; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Educational Problems
Keywords: Haptic education technology; Computer based simulation; Nursing education

STUDY DESIGN:
Intervention Model Description: The study is designed in a randomized controlled experimental type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After the theoretical lesson, the students in the experimental group were taken to the laboratory room where the 3D Systems Touch Haptic Simulator is located. The simulator has a choice of 45 minutes of full instruction, 5 minutes of haptic arm only, or the option. Since the preparation of the material in the full teaching method in the simulator takes a long time, these steps were removed to show similarity with the control group. The skill practice option for an average of 5-10 minutes where all steps of the Checklist for Teaching Urinary Catheterization Skill can be applied was used. Urinary catheterization with 3D Systems Touch Haptic Simulator was explained by 1 researcher who was responsible for the Fundamentals of Nursing course.
  Interventions: Device: 3D Systems Touch Haptic Simulator
- Control (No Intervention): After the theoretical lesson, the control group was taken to Fundamentals of Nursing Skill Laboratory. 1 researcher, who is responsible for the Fundamentals of Nursing, was explained on the Simple Urinary Catheterization Model by applying the steps of "Checklist for Teaching Urinary Catheterization Skills". The students were allowed to ask questions and the questions asked were answered. Then all the students in the control group were taken to an empty class. The two researchers prepared the necessary materials for the urinary catheterization skill practice in the same way in separate rooms. The doors were closed to keep the environment calm during the application. One student was taken to each laboratory rooms in order not to be affected by each other. While the student was practicing, both researchers filled in the Checklist for Teaching Urinary Catheterization Skills. Satisfaction Questionnaire was given to the student who completed the application and asked to fill it.

INTERVENTIONS:
Device: 3D Systems Touch Haptic Simulator — This simulator is computer-aided and allows us to see this application on the computer screen while practicing with a haptic arm. It gives real-like feedback in hand manipulations. The simulator has a choice of 45 minutes of full instruction, 5 minutes of haptic arm only, or the option.
  Arms: Intervention

SUMMARY:
Background: Haptic systems represent the highest level of computer based education technologies and enable students to learn at the highest level. These applications increase the student's focus as well as making the education non-monotonous and insuring teaching permanent by ensuring the active participation of the student.

Objective: The study was conducted to determine the effectiveness of using haptic technology in teaching urinary catheter application skill on the level of success and satisfaction about this skill.

DETAILED DESCRIPTION:
Method: This randomized-controlled experimental study was conducted with nursing students registered at a public university between December 2018 and March 2019. The sample of the study included 78 second grade students who gave consent after being informed about the aim of the study and who met the inclusion criteria. Control (n=39) and experimental (n=39) groups were determined through randomization using simple numbers table. Urinary catheterization application skill was taught with the standard curriculum (demonstration on the model) to the control group while it was taught with haptic-controlled computer based simulation technology to the experimental group. Data were collected using "Structured Student Introduction Form," "Skill Checklist for Teaching Urinary Catheterization Skill" and "Questionnaire for Satisfaction with Training Methods."

ELIGIBILITY:
Inclusion Criteria:

* being 18 years and over,
* enrolling for the first time in Fundamentals of Nursing course,
* participating in the study completely
* volunteering to participate

Exclusion Criteria:

* being a graduate of Health Vocational High School

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Urinary Catheterization Skill Score | through study completion, an average of 4 year
  The 25-item checklist prepared by the researchers based on the literature includes the application steps of urinary catheterization skill
Satisfaction Questionnaire | through study completion, an average of 2 year
  The survey consists of 16 statements and the participants were asked to give a score for each instruction method on a five-item Likert-type scale between 1 and 5 (1-absolutely not agree, 5-absolutely agree). It is found that as the scale score average increases, students' satisfaction with the educational method increases, and as the scale score average decreases, their satisfaction with the education method decreases. In the evaluation of the scale, students are given a minimum of 16 and a maximum of 80 points for their satisfaction with their educational methods.

CONTACTS AND LOCATIONS:
Overall Officials: Demet İnangil, Dr, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozturk D, Dinc L. Effect of web-based education on nursing students' urinary catheterization knowledge and skills. Nurse Educ Today. 2014 May;34(5):802-8. doi: 10.1016/j.nedt.2013.08.007. Epub 2013 Aug 20. PMID 24011752
- [Background] Jung EY, Park DK, Lee YH, Jo HS, Lim YS, Park RW. Evaluation of practical exercises using an intravenous simulator incorporating virtual reality and haptics device technologies. Nurse Educ Today. 2012 May;32(4):458-63. doi: 10.1016/j.nedt.2011.05.012. Epub 2011 Jun 12. PMID 21664014